CLINICAL TRIAL: NCT00669812
Title: A Phase II Evaluation of High Dose Chemotherapy and Autologous Stem Cell Transplantation for Intestinal T-cell Lymphomas
Brief Title: High-Dose Chemotherapy Given Together With Peripheral Blood Stem Cell Transplant in Treating Patients With Intestinal T-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593564; CRUK-2005-003906-27; CRUK-BRD/05/93
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: small intestine lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Carmustine; Cyclophosphamide; Cytarabine; Doxorubicin; Epirubicin; Etoposide; Ifosfamide; Melphalan; Methotrexate; Prednisolone; Vincristine; Biopsy; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Drug: methotrexate
Drug: prednisolone
Drug: vincristine sulfate
Procedure: autologous hematopoietic stem cell transplantation
Procedure: biopsy
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or by killing them. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This phase II trial is studying high-dose chemotherapy given together with peripheral blood stem cell transplant in treating patients with intestinal T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy and toxicity of intensive high-dose chemotherapy (alternating I'VE regimen and intermediate-dose methotrexate) followed by autologous peripheral blood stem cell transplantation for treatment of patients with intestinal T-cell lymphoma.

Secondary

* To assess the toxicity of the regimen in a large population of these patients.
* To provide a coordinated approach to the treatment of these patients.
* To register patients unfit for the protocol chemotherapy into the pathological part of the study.

OUTLINE: This is a multicenter study

* Chemotherapy: Patients receive CHOP chemotherapy comprising cyclophosphamide IV over 15 minutes, doxorubicin hydrochloride IV, and vincristine IV on day 1. Patients also receive oral prednisolone on days 1-5.

After recovering from CHOP chemotherapy, patients receive I'VE chemotherapy comprising epirubicin hydrochloride IV on day 1 and etoposide IV over 2 hours and ifosfamide IV continuously on days 21-23. Patients also receive methotrexate IV over 24 hours on day 21. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

* Consolidation therapy: On day 77, stem cells are collected from patients if the marrow is clear of disease. After completion of chemotherapy, patients in complete remission receive carmustine IV on day 105, cytarabine IV and etoposide IV on days 106-109, and melphalan IV on day 110. These patients undergo autologous peripheral blood stem cell transplantation on day 112.

Prior to study treatment, patients undergo a biopsy of the gut to confirm diagnosis and a blood sample is taken. Both blood and tissue samples may be used for further studies.

After recovery from treatment, patients are followed monthly for 4 months, then bimonthly for 1 year, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly confirmed diagnosis of intestinal T-cell lymphoma/ enteropathy-type T-cell lymphoma according to the following WHO classifications:

  * Usual phenotype CD3-, CD7-positive; CD5-, CD4-, CD8-negative; or CD30-positive
* Complete surgical resection allowed

PATIENT CHARACTERISTICS:

* Unsupported neutrophils ≥ 1,500/mm^3 unless attributed to lymphomatous bone marrow infiltration
* Unsupported platelets ≥ 100,000/mm^3 unless attributed to lymphomatous bone marrow infiltration
* Creatinine clearance ≥ 50 mL/min
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Left ventricular ejection fraction ≥ 50%
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* Patients with any serious concomitant medical or psychiatric condition that would preclude them tolerating the planned treatment should be entered into the registration study only
* No known hepatitis B, hepatitis C, or HIV positivity
* No active uncontrolled cardiovascular disease
* No abnormal EKG if there is a previous history of cardiac problems
* No other severe impairment of cardiac function
* No active malignancy within the past 5 years except cervical intraepithelial neoplasia or localized skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior diagnostic or emergency surgical procedures allowed
* More than 5 years since prior treatment for malignancy
* No prior chemotherapy or radiotherapy for treatment of lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Survival at 1 year

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lennard, Principal Investigator — Sir James Spence Institute of Child Health at Royal Victoria Infirmary
Locations (1):
- Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England, United Kingdom

REFERENCES:
- [Derived] Phillips EH, Lannon MM, Lopes A, Chadwick H, Jones G, Sieniawski M, Davies A, Wood K, Clifton-Hadley L, Smith P, Lawrie A, Chadwick N, Lennard AL. High-dose chemotherapy and autologous stem cell transplantation in enteropathy-associated and other aggressive T-cell lymphomas: a UK NCRI/Cancer Research UK Phase II Study. Bone Marrow Transplant. 2019 Mar;54(3):465-468. doi: 10.1038/s41409-018-0294-2. Epub 2018 Aug 13. No abstract available. PMID 30104718